CLINICAL TRIAL: NCT03280446
Title: Evaluation Using Intragen Fractional Radiofrequency With NeuViVa for the Treatment of Vaginal Laxity and Urogynecology Symptoms.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SHERRY Thomas (Other)
Responsible Party: Sponsor-Investigator, SHERRY Thomas, Sherry Thomas, MD, MPH, The American Association of Female Pelvic Medicine Specialists, Inc.
Organization: The American Association of Female Pelvic Medicine Specialists, Inc. (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IG-VL-101
Record Dates: First submitted 2017-09-01; First posted 2017-09-12 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Vaginal Laxity; Urinary Incontinence; Sexual Dysfunction
MeSH Terms: conditions — Urinary Incontinence; Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- 30 pre-menopause and post-menopause women (Experimental): Thirty healthy women with mild to moderate pelvic prolapse above the ages of 18 seeking treatment for vaginal laxity
  Interventions: Device: Intragen fractional radiofrequency with NeuViVa

INTERVENTIONS:
Device: Intragen fractional radiofrequency with NeuViVa — The Transcutaneous Fractional Radiofrequency Device (TFRF) is a minimal risk device that is currently cleared by the FDA K142833.The device uses a non-invasive, transepithelial treatment probe to elevate epithelial tissue temperatures to 40-45 oC for the purpose of promoting tissue contracture. Real-time tissue impedance monitoring will be carried out using the treatment probe.

SUMMARY:
This study will evaluate the clinical efficacy of a Transcutaneous Fractional Radiofrequency Device (TFRF) for the treatment of vaginal laxity (VL) and urogynecological symptoms.

DETAILED DESCRIPTION:
A total of thirty (30) subjects will be enrolled and assigned to a single treatment arm, receiving active treatment clinic, with the visits consisting of three (3) treatment administrations and post-procedure visits days 30, 180 and 360. Pre-menopausal and post-menopausal women between ages over 18, vaginal delivery, with up to moderate pelvic prolapse 2 cm past the hymen, and self-reported vaginal laxity score of "very loose", moderately loose", or "slightly loose" as defined by theVaginal Laxity Questionnaire (VLQ) will be evaluated and enrolled after having met all inclusion and exclusion criteria.

The treatment administration phase will consist of three (3) treatments,delivered approximately on-month apart. Subjects will be placed on the treatment table in the dorsal lithotomy position. The monopolar return pad will be placed on the subject buttock and to the RF generator.Coupling fluid will be used as a lubricant and will be reapplied throughout the treatment as needed. The treatment area is approximately 20+ cm2 and consist of the outside perineum and entire vaginal circumference along the length of the vagina to include the apex. For treatment of the labia majora, the treatment tip will be applied across the entire anatomical region. The treatment tip is applied to the perineum bilaterally from the lowest edge of the mons pubis to the perineal body and laterally to the crural folds to achieve vulvar and perineal temperatures of between 40-45 degrees celsius for approximately 5 minutes or more of total heat time per area. The labia majora and perineal areas will take approximately 10-15 minutes to complete. This is followed by treating the epithelial surface of the vaginal opening and advancing to the length of the vaginal canal with the treatment occurring along the vaginal walls, floor, and ceiling. The entire vaginal area will be treated in a circumferential area by delivering the RF in a systematic fashion at 5 separate delivery position starting the most distal portion of the vagina. The probe is slowly retracted at 1 cm intervals and circumferentially delivered again at 5 positions on another circumferentially manner moving the probe clockwise or counter clockwise or counter clockwise. To include the entire length of the urethra and bladder will be included in the treatment. Total vaginal treatment time will be 15-20 minutes. Safety measures will include monitoring of adverse events including pain or burns or infections during and after the procedure. Evaluations will be conducted with the visits at days 30, 90 and 150 days post-procedure.

During and after treatment administration, subjects will be asked to assess the self- reported pain experience using a 10 scale VAS, with "0" being no pain and "10" being the worst pain imaginable. Descriptive statistics will be generated on all demographic, medical history, and physical examination findings including means and standard deviations, for continuous, and frequencies and percentages for categorical variables.

ELIGIBILITY:
Inclusion Criteria:

Healthy female adult subjects presenting, clinically, with VL, and has expressed interest in treatment will be considered eligible for the study. Enrollment of subject will depend on meeting the following criteria:

* Voluntarily signed informed consent form
* Ages ≥ 18
* Completed urine pregnancy examination with negative result if premenopausal
* Self-reported perceptions of vaginal laxity deﬁned as "very loose," "moderately loose," or slightly loose" on the Vaginal Laxity Questionnaire.
* Up to Baden-Walker Grade 2 or Stage 2 Pelvic Organ Prolapse (≤ 1 cm past hymen)
* Papanicolaou smear cytology within 36 months prior to treatment showing no dysplasia
* Subject willing to take valacyclovir at 100 mg PO q12h x 3 for history recurrent episode of HSV
* or 1000mg PO q daily x 5 days

Exclusion Criteria:

* Baden-Walker System Severe pelvic prolapse (≥ Stage 3); Pelvic organ prolapse up to

  1 cm beyond the hymenal ring.
* Active STD (e.g. genital herpes, condylomata)
* Body mass index ≥ 35
* Previous reconstructive vaginal surgery, vaginal lasers, or vaginal injections of fat or fillers within 6 months.
* Current urinary tract infection
* Actively participating in, or planning on participating in, pelvic floor muscle strengthening exercises.
* Presence of pacemaker, AICD, or other electrical health maintenance device.
* Immunosuppression (pathological or medication induced, such as steroids, methotrexate) inﬂammatory drugs on a chronic basis (e.g., ibuprofen, aspirin and steroids) that can affect collagen or healing. Subject may qualify if willingly fulﬁlls a 30-day washout period of such drugs prior to treatment.They were using anti-inﬂammatory drugs on a chronic basis (e.g., ibuprofen, aspirin and steroids) that can affect collagen or healing. Subject may qualify if willingly fulﬁlls a 30 days washout period of such drugs prior to treatment.

Those with clinically signiﬁcant anxiety or depression that may prohibit completion of treatments and/or suffering a medical problem that might interfere with wound healing.

• All subjects on oral contraceptives prior to enrollment are encouraged to take these throughout the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-08-23 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of transcutaneous Fractional Radiofrequency Device (TFRF) for the treatment of vaginal laxity using the vaginal laxity questionnaire (VLQ). | 12 month
  The primary outcome measure is the mean change in the severity of the vaginal Laxity (VL) and in female Sexual Function Inventory (FSFI) by using VLQ, assessment and visual analog scale compared to base line.

SECONDARY OUTCOMES:
To evaluate the efficacy of transcutaneous Fractional Radiofrequency Device (TFRF) for the treatment of urogynecological symptoms. | 12 month
  To seasures improvement in subject sexual satisfaction and Urogynecological symptoms using sexual satisfaction Questionnaire (SSQ) and GRA (Global Response Assessment)

CONTACTS AND LOCATIONS:
Locations (1):
- The American Association of Female Pelvic Medicine Specialists, Inc., Agoura Hills, California, United States

IPD SHARING:
Plan to Share IPD: Undecided